CLINICAL TRIAL: NCT06477978
Title: The Prevalence of Sarcopenia in a Cohort of Patients With End Stage Kidney Disease on Haemodialysis Patients and Its Correlation With Mortality
Brief Title: The Prevalence of Sarcopenia in a Cohort of Haemodialysis Patients and Its Correlation With Mortality
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, Tarek Samy Abdelaziz, Associate professor of Internal medicine and nephrology, Kasr El Aini Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MD-119-2020
Record Dates: First submitted 2024-06-20; First posted 2024-06-27 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: End-stage Kidney Disease; End-stage Renal Disease; Dialysis Dependent Chronic Kidney Disease; Sarcopenia
Keywords: sarcopenia; end stage renal disease; end stage kidney disease; dialysis dependent end stage renal disease
MeSH Terms: conditions — Kidney Failure, Chronic; Sarcopenia

STUDY DESIGN:
Intervention Model Description: This is cohort prospective study of end stage kidney disease patients on hemodialysis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- End stage kidney disease patient on maintenance hemodialysis (Other): All patient that have been recruited with have the lean body mass index measured sing the Bio-impedance analysis ( BIA )
  Interventions: Diagnostic Test: Hand grip function testing

INTERVENTIONS:
Diagnostic Test: Hand grip function testing — The use of Bio-impedance to measure the skeletal muscle mass
  Other Names: Measuring skeletal body mass using bio-impedance analysis ( BIA)

SUMMARY:
The study aims to explore the correlation between the prevalence of sarcopenia and one year mortality amongst patients on maintenance hemodialysis

DETAILED DESCRIPTION:
In our study , we aim to explore the correlation between the prevalence of sarcopenia and one year mortality among patients on maintenance hemodialysis The lean muscle mass was measured using bio-impedance analysis (BIA ). The hand-grip test was used to measure the function .

Sarcopenia was defined using European Working Group on Sarcopenia in Older people (EWGSOP) definition which involves reduced muscle function and reduced muscle mass

ELIGIBILITY:
Inclusion Criteria:

* Patients with End stage kidney disease on maintenance dialysis

Exclusion Criteria:

* unable to consent or terminal malignancy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2021-02-15 (Actual); Primary Completion 2022-05-13 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
One year mortality | One year
  All cause mortality of patients with end stage kidney disease on hemodialysis

CONTACTS AND LOCATIONS:
Overall Officials: Tarek Abdelaziz, PhD, Principal Investigator — Kasr El Aini Hospital
Locations (1):
- Kasr Alainy University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No
Upon reasonable request